CLINICAL TRIAL: NCT03115671
Title: An Open-label Pilot Study on the Efficacy of Phosphatidylserine-Omega 3 (Vayarin) in Pediatric Patients Diagnosed With Autism and Comorbid Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Efficacy Study of Vayarin in Children With Autism and Comorbid Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Mental Health, Singapore (Other)
Responsible Party: Principal Investigator, Dr Sung Min, Senior Consultant, Psychiatrist, Institute of Mental Health, Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DSRB A/16/01120; CTC 1600529 (Other: Health Sciences Authority)
Record Dates: First submitted 2017-04-12; First posted 2017-04-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Autism Spectrum Disorder; Attention Deficit Hyperactivity Disorder
Keywords: Phosphatidylserine; Omega-3
MeSH Terms: conditions — Autism Spectrum Disorder; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Clinicians conducting the study assessments and teachers who will be providing feedback will be blinded to the study arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Each child participant in the Intervention group will be taking 4 capsules of Vayarin per day for 3 months. Each capsule contains 167mg Lipirinen, providing 75mg Phosphatidylserine (PS), 21.5mg EPA and 8.5mg DHA. This gives a daily dosage of 300mg PS and 120mg EPA/DHA. They may continue their treatment as usual provided there is no change in medication and intervention during the trial.
  Interventions: Dietary Supplement: Vayarin
- Control (No Intervention): Participants in the Control group will not be given Vayarin. They may continue their treatment as usual provided there is no change in medication and intervention during the trial.

INTERVENTIONS:
Dietary Supplement: Vayarin — Vayarin capsule
  Other Names: Phosphatidylserine-omega-3 (Lipirinen)
  Arms: Intervention

SUMMARY:
This research study is carried out to examine the effects of Phosphatidylserine-Omega 3 supplements (i.e., Vayarin) among children with Autism Spectrum Disorder (ASD) and ADHD. Participants will be randomised either to receive the Vayarin treatment (Intervention group) or to a Control group.

DETAILED DESCRIPTION:
There has been growing interest in the role of supplements such as omega-3 polyunsaturated fatty acids (n-3 PUFAs) in ADHD and ASD. Two of the primary n-3 PUFAs are eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), which are critical to brain development and are usually obtained through our diets. Increasing evidence has shown that children with ASD and/or ADHD have lower overall blood n-3 PUFAs levels than typically developing children (Parletta, Niyonsenga & Duff, 2016). Therefore, many studies have been conducted to examine the effectiveness of n-3 PUFAs supplementation among these two populations. While these supplements were found to have small but reliable benefit on ADHD symptoms (Hawkey & Nigg, 2014), there is limited evidence to support the use of n-3 PUFAs in clinical practice for the treatment of behavioural symptoms in children with ASD (James, Montgomery & Williams, 2011; Roux, 2015). Such inconsistencies give rise to the exploration of other alternatives in administering n-3 PUFAs.

Phosphatidylserine (PS), an acidic phospholipid (PL) molecule, comprises of a glycerol backbone esterified to the hydroxyl group of the amino acid serine via a phosphate group and to two fatty acids moiety (Manor et al., 2012). It plays a key role in the functioning of neuron membranes and may enhance the bioavailability of PUFAs. Administration of PL containing omega-3 PUFAs showed greater improvement in visual sustained attention performance among school children with ADHD, as compared to placebo and fish oil groups (Vaisman et al., 2008). Similarly, another study also suggested the benefits of PS-Omega3 (i.e., Vayarin) in reducing ADHD symptoms (Manor et al., 2012). This supplementation is shown to be generally safe and well-tolerated (Manor et al., 2013).

Nevertheless, these studies were conducted among children with ADHD. Given that n-3 PUFAs are commonly used by children with comorbid ASD and ADHD, there is a need to examine whether similar effects can be observed in this population. The goal of our present study is to examine the effect of PS-Omega3 supplement among children with comorbid ASD and ADHD. The safety and tolerability will also be assessed in this pilot trial.

ELIGIBILITY:
Inclusion Criteria:

* Between the age of 6 and 12 years old inclusive.
* Meets diagnostic criteria for ASD, based on Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5), and/or equivalent diagnosis based on Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR).
* Meets diagnostic criteria for ADHD (hyperactive/inattentive/combined subtype), based on Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5).
* Potential participants who are on stimulatory prescriptions should have no dose change 1 month prior to study initiation and throughout the study.
* Potential participants who are on other omega supplements to stop the supplements prior to the initiation and throughout the study.
* Potential participants who are on behavioural interventions should have no change in frequency or treatment plan 1 month prior to study initiation and throughout the study.

Exclusion Criteria:

* Girls who have reached menarche and presented with 3 previous regular menstrual cycles to minimize risk of adverse side effects.
* Change in dosage of psychiatric pharmacotherapy or other medications that have central nervous system effects or that affect performance, e.g., antidepressants (e.g. SSRIs, SNRIs), antipsychotics, adrenergic blockers, decongestant or sympathomimetics, anticonvulsants, mood stabilizers, melatonin, and sedating anti-histamines, or lithium carbonate 1 month before study initiation and throughout the study phase.
* Patients that would be contraindicated for Aspirin and Warfarin treatment or present with known allergic reactions or sensitivity to marine, soy or corn products, or any other illness that the clinician determines may jeopardize patient's health.
* Patients with a known genetic syndrome which may complicate the presentation of ASD (e.g. Fragile X, William's Syndrome, Prader-Willi etc.) or presenting with suspected brain or central nervous system condition.
* Patients who present with symptoms of psychosis or high risk condition such as mood issues and suicide risk or present with history of physical, sexual or emotional abuse
* Patients who did not adhere to the study procedures

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Conners 3rd Edition - Parent | 12 weeks, assessed at baseline and week 12
  Changes from baseline to Week 12 on Conners 3rd Edition - Parent
Social Responsiveness Scale (SRS) | 12 weeks, assessed at baseline and week 12
  Changes from baseline to Week 12 on Social Responsiveness Scale (SRS)
Aberrant Behaviour Checklist (ABC) | 12 weeks, assessed at baseline and week 12
  Change from baseline to Week 12 on the Aberrant Behaviour Checklist (ABC), specifically on irritability subscale

SECONDARY OUTCOMES:
Physical examination and safety evaluation (PAERS) | 12 weeks, assessed at baseline, week 6 and week 12
  Assessments of related side effects and adverse events of the supplements based on physical examination and safety evaluation (as measured by PAERS) at baseline, Week 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Min Sung, Dr, Principal Investigator — Institute of Mental Health, Singapore
Locations (1):
- Child Guidance Clinic, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manor I, Magen A, Keidar D, Rosen S, Tasker H, Cohen T, Richter Y, Zaaroor-Regev D, Manor Y, Weizman A. The effect of phosphatidylserine containing Omega3 fatty-acids on attention-deficit hyperactivity disorder symptoms in children: a double-blind placebo-controlled trial, followed by an open-label extension. Eur Psychiatry. 2012 Jul;27(5):335-42. doi: 10.1016/j.eurpsy.2011.05.004. Epub 2011 Jul 31. PMID 21807480
- [Background] Manor I, Magen A, Keidar D, Rosen S, Tasker H, Cohen T, Richter Y, Zaaroor-Regev D, Manor Y, Weizman A. Safety of phosphatidylserine containing omega3 fatty acids in ADHD children: a double-blind placebo-controlled trial followed by an open-label extension. Eur Psychiatry. 2013 Aug;28(6):386-91. doi: 10.1016/j.eurpsy.2012.11.001. Epub 2013 Jan 9. PMID 23312676
- [Background] Vaisman N, Kaysar N, Zaruk-Adasha Y, Pelled D, Brichon G, Zwingelstein G, Bodennec J. Correlation between changes in blood fatty acid composition and visual sustained attention performance in children with inattention: effect of dietary n-3 fatty acids containing phospholipids. Am J Clin Nutr. 2008 May;87(5):1170-80. doi: 10.1093/ajcn/87.5.1170. PMID 18469236